CLINICAL TRIAL: NCT01845844
Title: Ranibizumab For Persistent Diabetic Macular Edema After Bevacizumab (ROTATE Trial)
Brief Title: Ranibizumab For Persistent Diabetic Macular Edema After Bevacizumab
Acronym: ROTATE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast Retina Center, Georgia (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Dennis M. Marcus, M.D., Dr. Dennis M. Marcus Principal Investigator, Southeast Retina Center, Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28713
Record Dates: First submitted 2013-04-02; First posted 2013-05-03 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab 0.3mg (12 months) (Experimental): Intravitreal injection of ranibizumab 0.3mg/0.05cc
  Interventions: Drug: Ranibizumab 0.3mg/0.05cc
- Ranibizumab 0.3mg (6 months) (Active Comparator): Intravitreal injection of ranibizumab 0.3mg/0.05cc
  Interventions: Drug: Ranibizumab 0.3mg/0.05cc

INTERVENTIONS:
Drug: Ranibizumab 0.3mg/0.05cc — Group A (Arm A) will receive monthly 0.3mg/0.05cc intravitreal injections for 12 consecutive months.
  Group B (Arm B) will receive monthly 0.3mg/0.05cc intravitreal injections for the first six months and then PRN for the remaining 6 months per protocol specified criteria.
  Other Names: Lucentis

SUMMARY:
This is an open-label, Phase I/II study of Intravitreally administered 0.3mg ranibizumab in subjects with persistent Diabetic Macular Edema (DME) after recent and frequent bevacizumab (at least 2 bevacizumab intravitreal injections within 2 months prior to enrollment and at least 6 bevacizumab injections within 9 months of enrollment).

DETAILED DESCRIPTION:
30 eyes will be randomized in a 1:2 ratio (Group A= 10 patients; Group B= 20 patients) Group A: ("monthly group")- Consented patient with enrolled eye will receive 12 monthly required injections of 0.3mg ranibizumab over 1 year OR Group B: ("As needed (PRN) Group")- Consented patient with enrolled eye will receive 6 monthly required injections of 0.3mg ranibizumab for 6 months, followed by as needed (PRN) dosing (required ranibizumab if DME persistent on Optical Coherence Tomography (OCT) and Early Treatment Diabetic Retina Study (ETDRS) Best Corrected Visual Acuity (BCVA) <20/20) for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* >=18 years
* Type I/II diabetes mellitus
* Central-involved DME in study eye (OCT CSF >=275um on Heidelberg Spectralis spectral domain OCT with evidence of intraretinal or subretinal fluid or cysts)
* Definite retinal thickening due to diabetic macular edema involving the center of the macula.
* Media clarity, pupillary dilation and individual cooperation for adequate fungus photography and fluorescein angiography.
* Visual Acuity score in study eye <=80 and >=20 (approximate Snellen equivalent 20/25 to 20/400).
* History of at least 6 intravitreal bevacizumab injections within the past 9 months and 2 intravitreal bevacizumab injections within the past 2 months.
* No history of an anti-VEGF treatment for DME in the past 3 weeks.
* No other DME treatment for DME, other than bevacizumab, in the study eye at any time in the past 3 months.
* No history of major ocular surgery in the study eye within prior 3 months or anticipated within the next six months following randomization.

Exclusion Criteria:

* Pregnancy or lactation
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another medical investigation or trial within 30 days of randomization
* Known allergy to ranibizumab
* Acute cardiovascular event requiring hospitalization within the past 3 months
* Systemic anti-VEGF or pro-VEGF treatment within 3 months prior to randomization or anticipated use during the study
* Macular edema is considered to be due to a cause other than DME
* An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from the resolution of macular edema
* History of intravitreal anti-vascular endothelial growth factor (anti-VEGF) agent other than bevacizumab within 9 months prior to randomization
* History of panretinal photocoagulation within 3 months prior to randomization or anticipated need for panretinal photocoagulation in the 6 months following randomization
* Yag capsulotomy performed within 1 month prior to randomization
* External ocular infection including conjunctivitis, significant blepharitis, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular and systemic adverse events will be compared between experimental and active comparator groups | 1 year
  Examples include worsened acuity of greater than 30 letters, retinal detachment, endophthalmitis, cataract progression, vitreous hemorrhage, new PDR or neovascularization of the iris or angle, incidence and severity of other adverse events, as identified by physical examination, subject reporting, and changes in vital signs and will include thromboembolic events, deaths and systemic serious adverse events
Severity of ocular and systemic adverse events will be compared between experimental and active comparator groups | 1 year
  Examples include worsened acuity of greater than 30 letters, retinal detachment, endophthalmitis, cataract progression, vitreous hemorrhage, new PDR or neovascularization of the iris or angle, incidence and severity of other adverse events, as identified by physical examination, subject reporting, and changes in vital signs and will include thromboembolic events, deaths and systemic serious adverse events

SECONDARY OUTCOMES:
Efficacy of monthly and monthly followed by PRN dosing of 0.3 mg ranibizumab after persistent DME despite previous bevacizumab therapy | 1 year
  Examples include proportion of eyes with absence of fluorescein angiographic macular leakage at 12 months; proportion of eyes with unchanged, worsened, or improved fluorescein angiographic macular leakage from baseline at 1, 6 and 12 months; proportion of eyes with unchanged, worsened, or improved fundus photographic DME appearance from baseline at 1, 6 and 12 months; proportion of eyes with new vitreous hemorrhage or traction retinal detachment secondary to Proliferative Diabetic Retinopathy (PDR); proportion of eyes with progression from baseline Non-proliferative Diabetic Retinopathy (NPDR) to PDR

OTHER OUTCOMES:
Mean BCVA letter score | Baseline, 1, 3, 6, 9, and 12 months
  ◦Mean BCVA letter changes from baseline at 1, 3, 6, 9 and 12 months
Mean OCT CSF thickness and macular volume | Baseline, 1, 3, 6, 9, and 12 months
  OCT Central Subfield (CSF) thickness and macular volume mean changes from baseline at 1, 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dennis M Marcus, M.D., Study Director — Southeast Retina Center
Locations (1):
- Southeast Retina Center, PC, Augusta, Georgia, United States